CLINICAL TRIAL: NCT01180088
Title: Effectiveness of Routine Application Of Anterior Approach During Right Hepatectomy: A Randomized Trial
Brief Title: Effectiveness of Routine Application Of Anterior Approach During Right Hepatectomy
Acronym: AA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera Ordine Mauriziano di Torino (Other)
Responsible Party: Lorenzo Capussotti MD, Azienda Ospedaliera Ordine Mauriziano di Torino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AA001
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Liver Neoplasm
Keywords: LIVER TUMOURS
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ANTERIOR APPROACH (Experimental): SURGICAL TECHNIQUE
  Interventions: Procedure: RIGHT HEPATECTOMY WITH CLASSIC APPROACH

INTERVENTIONS:
Procedure: RIGHT HEPATECTOMY WITH CLASSIC APPROACH — The right portal branch and the right branch of the hepatic artery were identified, dissected and divided. Extraparenchymal ligation of pedicles for Sg4 was performed in case of extended right hepatectomy. The falciform and the right triangular ligaments were sectioned and the right liver up to the retrohepatic vena cava was totally mobilized by section and sutures of the accessory right hepatic veins. The right hepatic vein was controlled in an extrahepatic plane and encircled with a tape. At the end of parenchymal transection right hepatic vein was sectioned with endovascular stapler. The right bile duct and middle hepatic vein (in case of extended right hepatectomy) were divided intraparenchymally
  Other Names: Right Hepatectomy

SUMMARY:
The aim of this study was to evaluated the advantages of routine application of the anterior approach in patients scheduled to right hepatectomy or extended right hepatectomy, without infiltration of segment 1, inferior vena cava or main bile duct.

DETAILED DESCRIPTION:
Mobilization of the liver during right hepatectomy with classic approach is performed before parenchymal transection. In this phase severe bleeding may occur due to laceration of the inferior vena cava (IVC) wall, rupture or ligation falling off the hepatic short vein (HSV) or bleeding from the right liver attachments. Besides, the twisting of the portal pedicle during mobilization can render the left hepatic lobe ischemic for transient interruption of the hepatopetal flow. These events are more frequent in case of large hepatic lesions (mainly HCC) that involves surrounding structures (such as diaphragm). Two of the most important factors that affect the postoperative course of patients undergoing liver resections are indeed intraoperative bleeding and postoperative liver dysfunction. For these reasons Lai et al proposed anterior approach as alternative to classic right hepatectomy. In this case liver mobilization is performed only at the end of parenchymal transection, when all vascular connections are already interrupted. Liu et al published the results of a retrospective study in which 54 patients with, right sided HCC greater than 5 cm underwent right hepatectomy using the anterior approach technique. The anterior approach group had significantly less intraoperative blood loss, less need of blood transfusion and a lower hospital mortality rate. The same group reported results of a prospective randomized controlled study analyzing 120 patients with large (>5 cm) right liver HCC. The overall operative blood loss, morbidity, and duration of hospital stay were comparable in both groups. However, a higher number of patients in classic approach group experienced mayor operative blood loss (> 2000 cc) and required blood transfusions (8.3% vs. 28.3%).

ELIGIBILITY:
Inclusion Criteria:

* patients between 18 and 80 years
* patients scheduled to right hepatectomy or extended right hepatectomy
* the future remnant liver (FRL) ≥ 25% in patients with a normal liver or ≥ 30% in those with chronic liver disease
* indocyanine green retention rate (ICG) at 15 minutes ≤ 10% in cirrhotic patients

Exclusion Criteria:

* resection of S1
* resection of bile duct
* infiltration of inferior vena cava
* America Society of Anesthesiologists (ASA) grade IV
* Emergency surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-09 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
OVERALL BLOOD LOSS | UP TO 7 DAYS

SECONDARY OUTCOMES:
BLOOD TRANSFUSION RATE | WITHIN 24 HOURS

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Capussotti, MD, Principal Investigator — Ospedale Mauriziano di Torino
Locations (1):
- Ospedale Mauriziano di Torino, Turin, Italy

REFERENCES:
- [Background] Lai EC, Fan ST, Lo CM, Chu KM, Liu CL. Anterior approach for difficult major right hepatectomy. World J Surg. 1996 Mar-Apr;20(3):314-7; discussion 318. doi: 10.1007/s002689900050. PMID 8661837
- [Background] Liu CL, Fan ST, Cheung ST, Lo CM, Ng IO, Wong J. Anterior approach versus conventional approach right hepatic resection for large hepatocellular carcinoma: a prospective randomized controlled study. Ann Surg. 2006 Aug;244(2):194-203. doi: 10.1097/01.sla.0000225095.18754.45. PMID 16858181
- [Background] Liu CL, Fan ST, Lo CM, Tung-Ping Poon R, Wong J. Anterior approach for major right hepatic resection for large hepatocellular carcinoma. Ann Surg. 2000 Jul;232(1):25-31. doi: 10.1097/00000658-200007000-00004. PMID 10862191
- [Derived] Capussotti L, Ferrero A, Russolillo N, Langella S, Lo Tesoriere R, Vigano L. Routine anterior approach during right hepatectomy: results of a prospective randomised controlled trial. J Gastrointest Surg. 2012 Jul;16(7):1324-32. doi: 10.1007/s11605-012-1894-6. Epub 2012 May 9. PMID 22570073